CLINICAL TRIAL: NCT06423391
Title: A Multimodal Manual Therapy-Based Intervention for People With Painful Diabetic Neuropathy: Feasibility of a Randomised Controlled Efficacy Trial
Brief Title: Multimodal Intervention for Painful Diabetic Neuropathy: NeuOst Feasibility Trial
Acronym: NeuOst
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Osteopathy (Other)
Collaborators: Imperial College London (Other); King's College London (Other); University of Oxford (Other); Universität Münster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NeuOst feasib V 1.0 March 2024
Record Dates: First submitted 2024-05-09; First posted 2024-05-21 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-05

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: feasibility study of a single-site parallel three-armed participant-blinded controlled randomised trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The following stakeholders will be blinded to participants' group allocation in the test intervention and control intervention groups. Allocation to the Usual Care group will not be concealed from staff or participants, except for the trial statistician:
  * Trial participants (except in usual care arm)
  * Clinical support and administration staff
  * Outcome assessors (collecting data at end-of-treatment and follow-up)
  * Trial statistician
    * Provider blinding will not be possible as providers will have to actively deliver both the test and the control intervention. However, extensive pre-trial training and supervision during the trial will ensure that providers understand the purpose of the control intervention and are supported to deliver it with high fidelity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tested intervention (NeuOst treatment) (Experimental): The tested treatment is a manual therapy-based intervention, drawing on core manual therapy components and integrating psychologically informed approaches to pain management and elements from diabetes education, foot care, and exercise rehabilitation. This intervention is called 'Augmented manual therapy for people with painful diabetic neuropathy', or NeuOst. NeuOst components will be taught to fully qualified UK-registered osteopaths who then deliver the intervention according to a treatment manual in 1:1 appointments, lasting 45-60 minutes each (90 mins first appointment). Up to 5 treatment sessions will be provided per patient, at weekly intervals and at maximum over 10n weeks.
  The treatment manual specifies obligatory and optional elements for each of the 5 study treatment sessions. Exercise components will be rehearsed in the clinic with providers. Participants will then be encouraged to complete a progressive home-exercise programme according to the manual.
  Interventions: Other: NeuOst
- Control intervention (Sham Comparator): The objectives of the control intervention are to replicate the contextual elements of the test intervention (to test efficacy), and to blind participants to group allocation. Trial providers will be trained in its delivery. As per CoPPS guidance, the control intervention will resemble the tested intervention in all aspects but for the components whose effect the trial is designed to study. These excluded components of interest, and their respective adaptations in the control intervention, are specified in the detailed pre-registered protocol.
  Control intervention components will be taught to fully qualified UK-registered osteopaths who then deliver the intervention according to a treatment manual in 1:1 appointments, lasting 45-60 minutes each (90 mins first appointment). Up to 5 treatment sessions will be provided per patient, at weekly intervals and at maximum over 10 weeks.
  Interventions: Other: Control Intervention
- Usual care comparator (Other): Participants randomized to this study arm will only undergo baseline and follow-up assessments but will receive no further attention as part of this trial. As in all other trial arms, they are free to continue their usual medical care but will be encouraged to not change their analgesic regime or nonpharmacological management as far as possible.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: NeuOst — As above
  Arms: Tested intervention (NeuOst treatment)
Other: Control Intervention — As above
  Arms: Control intervention
Other: Usual Care — As above
  Other Names: Treatment as Usual
  Arms: Usual care comparator

SUMMARY:
This is the feasibility study of a single-site parallel three-armed participant-blinded controlled randomised efficacy trial of a 5-week course of the 'NeuOst treatment', compared to a designated control intervention, and to usual care only, for adults with pDPN.

DETAILED DESCRIPTION:
Eligible participants are adults diagnosed with diabetes and pDPN, as evaluated with clinical questionnaires during an initial telephone screening. Participants with foot ulcerations, amputations, and advanced organ failure are excluded. Twelve participants per arm (36 in total) will be recruited via social media, local print media, and a poster and leaflet campaign in relevant clinics.

Blocked randomisation will allocate participants in a 1:1:1 ratio, using permuted block sizes. The test intervention consists of five weekly 1-hour sessions of semi-standardised augmented manual therapy with a specifically trained provider (NeuOst), in addition to participants' continued usual care. The control intervention will be specifically matched following current guidance, replicating the NeuOst intervention in all aspects except selected components which the study aims to investigate. Providers will be UK-registered osteopaths. Both test and control intervention were developed with extensive involvement of people with pDPN and practitioners. The third study arm will be a Usual Care (UC) group, consisting of baseline and follow-up assessments only. All trial participants can continue their usual care outside the trial, although participants will be asked to not alter their medication regimens or nonpharmacological management if possible.

An independent combined steering & data-monitoring committee (TSC/DMC) will monitor the trial throughout and include a stakeholder representative. Participants will be reimbursed for their travel expenses but not time. Screening and follow-up data collection will be conducted electronically or via the phone to minimise trial burden. The timepoints of follow-up are immediately after treatment completion, and at 8 and 16 weeks from randomisation.

Key methodological and reporting guidance for feasibility trials will be followed, and a protocol pre-registered. Ethical approval was obtained from the institutional Research Ethics Committee.

Feasibility of a definite trial will be judged according to pre-specified criteria regarding the primary feasibility outcomes following pre-specified progression rules: Recruitment, consent rates, treatment completion, retention rates, interventionist fidelity in treatment delivery, data completeness, treatment acceptability, blinding success, and adverse events. Secondary outcomes include measures of pain intensity, interference, and quality, sleep, quality of life, and fear of falling.

The sample size of 36 was a pragmatic decision based on available funding and the trial is not powered to detect meaningful differences in clinical outcomes. Analysis of feasibility outcomes will be largely descriptive. For clinical outcomes, a pre-specified blinded analysis will provide estimates of changes in clinical outcome measures and their variance, modelling differently sized confidence intervals and presenting them as forest plot with the MCID indicated. This information can then be used for sample size calculations for a potential full-scale trial. Qualitative data from interviews with volunteering participants and trial interventionists will provide further nuance for progression decisions or intervention refinement.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of diabetes mellitus (type 1 or type 2) as per patient self-report.
* Distal symmetrical peripheral neuropathy (defined as a score of ≥4 on the Michigan Neuropathy Screening Instrument (questionnaire part) (Herman et al., 2012)).
* Neuropathic pain as assessed by DN4 questionnaire (defined as a score of ≥3 of 7 self-reported items) (Spallone et al., 2012).
* Stable analgesic medication regimen for at least 3 weeks prior to anticipated study enrolment and no revision of regimen planned within the next 3 months.
* Stable attendance of out-of-study nonpharmacological therapies for neuropathic pain or professional exercise programmes (including gym classes and manual therapy) for at least 3 weeks prior to anticipated study enrolment and no revision of routine planned within the next 3 months.
* Participants capable of giving informed consent themselves.
* Participants able to speak, understand, and read English at conversational levels.
* Age: 18 and older.

Exclusion Criteria:

* Contraindications to manual therapy and conservative pain management (as determined by recruiting staff during screening calls or the trial provider at the initial or any other appointment; May include medical emergencies and suspected severe pathology, advanced osteoporosis, and active foot ulcerations)
* Past or scheduled amputations
* Advanced renal failure
* Recent physical trauma and suspected fracture
* Currently experiencing severe depressive or other current and severe psychopathology such as bipolar/psychosis, and/or presenting with active suicidal risk
* Carpal Tunnel Syndrome diagnosis or symptoms as the only source of neuropathic pain
* Unable or unwilling to provide consent for study participation
* Unable to attend in-person appointments at treatment site (for health reasons)
* Unable to attend in-person appointments at treatment site (for organisational reasons)
* Knowing other participants signed up to the study (to avoid group contamination)
* Concomitant participation in another clinical intervention study
* Changes in medication or physical activity programmes in the past 1 month or planned for the next 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Study Feasibility | 12 months from recruitment start
  Using pre-defined set of feasibility criteria, measuring recruitment, consent rates, treatment completion, retention rates, interventionist fidelity in treatment delivery, treatment acceptability, blinding success, data completeness, adverse events, and participant acceptability.

SECONDARY OUTCOMES:
Pain intensity (average in past week) | 1, 2, 3, 4, 5, 8, 16 weeks
  measured on the Brief Pain Inventory (Short Form)
Impact of Diabetic Neuropathic Pain | 5, 8, 16 weeks
  measured on the Diabetic Peripheral Neuropathic Pain Impact (DPNPI) measure
Neuropathy- and Foot Ulcer-Specific Quality of Life | 5, 8, 16 weeks
  Neuropathy- and foot ulcer-specific quality of life instrument (NeuroQoL)
Fear of Falling | 5, 8, 16 weeks
  Falls Efficacy Scale (FES-I, short form)

OTHER OUTCOMES:
Global Impression of Change | 5, 8, 16 weeks
  Patient's Global Impression of Change scale
Concomitant medication and intervention use | 5, 8, 16 weeks
  Concomitant medication and intervention use via self-reported questionnaire
Pain Bothersomeness | 1, 2, 3, 4, 5, 8, 16 weeks
  measured as number of days with 'bothersome' and 'intolerable' pain in past week
Pain Intolerability | 1, 2, 3, 4, 5, 8, 16 weeks
  measured as number of days with 'intolerable' pain in past week
Participant experiences | 16 weeks
  Participant feedback form and semi-structured interviews on NeuOst and trial-related aspects

CONTACTS AND LOCATIONS:
Overall Officials: David Hohenschurz-Schmidt, PhD, Principal Investigator — University College of Osteopathy / Imperial College London
Locations (1):
- University College of Osteopathy, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The sharing of trial data, specifically anonymised individual patient data and summary data, is permissible once the final report of all analyses specified in this report has been published in a scientific journal. External parties can request access to this dataset or the dataset may be shared on an online repository (OSF.io).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once the final report of all analyses specified in this report has been published in a scientific journal.
Access Criteria: Anyone can access
URL: https://osf.io/sbqce/

REFERENCES:
- [Derived] Hohenschurz-Schmidt D, Smith S, Schmid AB, Bright P, Draper-Rodi J, Evans MC, Kemp H, Esteves NK, Pigott E, Scott W, Vollert J, Williamson E, Pogatzki-Zahn EM, Vogel S. A multimodal intervention of manual therapy, exercise, and psychological management for painful diabetic neuropathy: intervention development and feasibility trial protocol. Pain Manag. 2025 Jul;15(7):387-399. doi: 10.1080/17581869.2025.2515010. Epub 2025 Jun 11. PMID 40495635
- See also: Full protocol (embargoed until Nov 2024) — https://osf.io/sbqce/
- See also: Study website — https://www.hsu.ac.uk/research/neuost/

DOCUMENTS (1):
  • Informed Consent Form (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT06423391/ICF_000.pdf